CLINICAL TRIAL: NCT04626700
Title: Thoracic Department, Chang Gung Memorial Hospital, Linko Main Branch
Brief Title: Comparison for Oral Negative Pressure Therapy and CPAP for OSA Under Sleep Endoscopy Assistance: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201802177A3
Record Dates: First submitted 2020-11-01; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: OSA; iNAP; DISE

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iNAP (Experimental)
  Interventions: Device: iNAP
- CPAP (Active Comparator)
  Interventions: Device: CPAP

INTERVENTIONS:
Device: iNAP — iNAP for the treatment of OSA
  Arms: iNAP
Device: CPAP — CPAP for the treatment of OSA
  Arms: CPAP

SUMMARY:
This is the study entitled "Comparison for oral negative pressure therapy and CPAP for OSA under sleep endoscopy assistance: A randomized controlled trial". CPAP is first line golden standard treatment for Obstructive sleep apnea (OSA). However, the overall CPAP compliance is poor. Recent study reveals that oral negative pressure therapy improves apnea severity in OSA patients with good compliance. However, no study is designed to compare oral negative pressure therapy and CPAP for OSA patients. In addition, the effect of oral negative pressure therapy for hypopharynx is unclear. Therefore, we will perform druginduced sleep endoscopy to evaluate upper airway obstruction of OSA patients before treatment. OSA patients will be assigned into oral negative pressure group or CPAP group for 2 months. Sleepiness, sleep quality, residual apnea severity and compliance will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate OSA

Exclusion Criteria:

* hypopharynx obstruction
* ASA classification of physical status)>3
* allergy toDexmedetomidine
* COPD stage IV
* Asthma with exacerbation
* severe CHF
* age < 18 year-old
* claustraphobia
* any reason : can not tolerate CPAP
* second or third degree AVB

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The Epworth Sleepiness Scale (ESS) | Change from Baseline ESS at 1 month
  lower ESS means better outcome
The Epworth Sleepiness Scale (ESS) | Change from Baseline ESS at 2 months
  lower ESS means better outcome
apnea-hypopnea index (AHI) | Change from Baseline AHI at 2 months
  lower AHI means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, MD, Study Chair — Institutional Review Board Chang Gung Medical Foundation
Locations (1):
- Division of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan